CLINICAL TRIAL: NCT06499909
Title: Hypnosis for the Management of Postoperative Pain Following Colectomies: a Single Centre Randomised Controlled Feasibility Trial
Brief Title: Hypnosis for Colectomies as Postoperative Pain Management
Acronym: Hypnopal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somerset NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 303418
Record Dates: First submitted 2024-06-11; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: to Evaluate the Effects of Clinical Hypnosis on Post-operative Pain, Following Colectomy Operations
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis (Experimental): Patient receives hypnosis treatment prior to surgery
  Interventions: Other: Hypnosis
- Normal care pathway (No Intervention): Patient will receive standard care

INTERVENTIONS:
Other: Hypnosis — The patient will receive a course of hypnosis
  Arms: Hypnosis

SUMMARY:
The present study intends to assess the feasibility, value and direction of conducting a future, full scale randomised controlled trial, to evaluate the effects of clinical hypnosis on post-operative pain, following colectomy operations.

Pain management in the postoperative setting presents a challenge as the development and severity of pain after surgery is dependent on different patient and procedural factors. Furthermore, pain after surgery is a major concern for patients, especially when it is undermanaged. When postoperative pain control is suboptimal it delays mobilisation, reduces oral food and fluid intake after surgery, and increases the risk of developing chronic pain and other complications. These factors have a negative impact on the patient recovery process, thus increasing the length of hospital stay and healthcare costs. Hypnosis is well recognised as having an effect in pain perception, it is a brief, easy to administer intervention making it a promising non-pharmacological intervention with the potential to help postoperative pain management in patients undergoing colectomies as well as reducing anxiety and emotional stress related to surgery, while also having a positive indirect effect on recovery times, which could lead to considerable cost-savings at organisational level.

The intervention will be delivered at Somerset NHS Foundation Trust by a designated Principal Investigator. Hypnosis sessions will be given face to face in a clinical consulting room and on the ward where the participants will be admitted after surgery. The study aims to enrol 40 participants, 20 for each arm, over 12 months, from Musgrove Park Hospital who will undergo elective colectomy surgery. Eligible participants would be adults 18 years or over, undergoing elective colectomy surgery. Participants must be able to provide a written informed consent and able to understand and communicate in English.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the study if they meet ALL of the following inclusion criteria

* Aged 18 years or over;
* Undergoing elective colectomy surgery (open and laparoscopic colectomies will be included).
* Patients that can provide written informed consent.
* Are able to understand and communicate in English.

Exclusion Criteria:

A patient meeting ANY of the following exclusion criteria at baseline will be excluded from participation:

* Emergency colectomies will be excluded due to the urgency of the intervention.
* Non English speakers.
* Patients with the following diagnosed mental health illness: personality disorders, psychosis or schizophrenia as hypnosis could aggravate these conditions.
* Patients that are already involved in other research studies and that could influence the results of the study.
* Any patient that is clinically unwell post-surgery with a National Early Warning Score (NEWS) of 5 or higher. NEWSscore is a tool developed for NHS England which improves the detection and response to clinical deterioration in adult patients and is a key element of patient safety and improving patient outcomes.
* Patients with deafness or difficulty hearing as this would be essential for this therapy to be effective.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
The effectiveness of hypnotic analgesia on post-operative pain after colectomies. | 365 days
  we are assessing the effectiveness of hypnosis on pain by using numeric pain scales to assess pain scores before and after hypnosis. This will then help us evaluate pain scores between groups and compare the before and after hypnosis scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Somerset NHS Foundation Trust, Taunton, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No